CLINICAL TRIAL: NCT06753435
Title: Development of the Premature Infant's Stress System. Focus on Parent-infant Co-regulation and Interaction
Brief Title: Co-regulation and Interaction in the NICU
Acronym: CORI
Status: Recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other)
Responsible Party: Principal Investigator, Evalotte Morelius, Professor, Linkoeping University
Other Study IDs: Dnr 2024-02916-01 CORI
Record Dates: First submitted 2024-12-12; First posted 2024-12-31 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Preterm
Keywords: Preterm infant; Stress system; Family
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva for analyse of cortisol and alpha-amylase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Families of preterm babies born at GA 30+0-34+6 enrolled in NICU

SUMMARY:
Preterm infants are exposed to multiple stressors each day, posing a risk of toxic stress that can impact their developing brains during a critical period of sensitivity. Elevated levels of the stress hormone cortisol can impede neuronal connectivity and communication, thereby increasing the likelihood of cognitive impairment and behavioural problems. Synchronized social-emotional mother-infant interaction holds promise in buffering stress reactivity and mitigating long-term stress effects.

Our previous research has shown that preterm infants exhibit higher baseline saliva cortisol levels than full-term infants, along with blunted cortisol reactivity to stressors, irregular cortisol circadian rhythms, and delayed cortisol co-regulation between mother and infant. Another potential stress marker is saliva alpha-amylase (α-amylase), which has garnered increasing interest in adult research. However, there remains a significant gap in the literature concerning saliva α-amylase as a stress marker in preterm infants, warranting further investigation. The overall aim is to study development and relationships between three systems of parent-infant synchrony in preterm infants and their parents and elucidate potential confounding factors for a synchronous correlation. This will be done in relation to standardised care procedures commonly performed in the neonatal intensive care unit.

This observational study will involve 35 families undergoing three video-recorded procedures in the NICU. Saliva will be collected from infants and both parents before and after each procedure so we can analyse co-regulation of cortisol and alpha-amylase. Parent-infant interaction will be analysed from the videos using validated scales.

This study will be the first to document biological co-regulation and social-emotional parent-infant interaction simultaneously involving preterm infants and both parents in the NICU setting. Such insights are pivotal for the future design and implementation of tailored nursing interventions aimed at early stress mitigation, thereby reducing the risk of stress-related consequences.

DETAILED DESCRIPTION:
This observational study adopts a correlational approach to investigate biological co-regulation and parent-infant interaction within families of preterm infants, utilizing a within-family design. Data collection occurs at multiple time points in the NICU, and at 6 and 12 months corrected age. To study parent-infant synchrony and co-regulation with both parents, both should be present and perform three diaper changes in three days. Two will be perforemd by the mother and one by the father. All occassions will be video recorded to study interaction and saliva will be collected before and after the procedure to study co-regulation in cortisol and alpha-amylase during baseline, reactivity and recocvery. At 6 and 12 months parents will respond to questionnaires regarding the child's behavior and development.

Sample size: A power calculation shows sample size of n=28 is sufficient, considering α (two-tailed) = 0.05, β = 0.20, and ICC = 0.5.To consider attrition, we paln to include 35 families.

ELIGIBILITY:
Inclusion Criteria:

* Swedish- or English-speaking parents aged over 18, born in Europe, and their infants born between gestational weeks 30+0 and 34+6.

Exclusion Criteria:

* Parents with conditions or taking medications affecting the hormone system. Additionally, infants with major malformations or complex care needs that impede interaction possibilities are excluded.

Min Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants born preterm between 30+0 and 34+6 weeks gestational age and their parents > 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Saliva cortisol correlation (co-regulation) within the triad (mother, father, infant) | GW 32 +/- 2 weeks
  Saliva will be collected from the infant and both parents before (baseline) and at 20 minutes (reactivity), and 40 minutes (recovery) after a diaper change performed three times in three days. Samples will be collected using swabs and stored frozen (-80C) until analysis. Cortisol will be analysed at Linköping University (LiU).
Saliva Alpha-amylase correlation (co-regulation) within the triad (mother, father, infant) | GW 32 +/- 2 weeks
  Saliva α-amylase will be collected from the infant and both parents before (baseline) and at 5 minutes (reactivity), 20 minutes (recovery) after a diaper change performed three times in three days. Samples will be collected using swabs and stored frozen (-80C) until analysis. α-amylase levels will be analysed at Linköping University (LiU).
Parent-infant emotional availability | GW 32 +/- 2 weeks
  All three diaper changes will be video recorded with both parents present and instructed to act as they normally would. Emotional availability will be evaluated from videos using the Emotional Availability Scales (EAS) by certified coders. EAS assesses dyadic and emotional qualities of parent-infant relationships across six sub-scales, with dimensions measured using a Likert-scale ranging from 1 to 7, higher scores indicate better emotional availability.
Parent-infant synchrony | GW 32 +/- 2 weeks
  All three diaper changes will be video recorded with both parents present and instructed to act as they normally would. Parent-infant synchrony will be assessed from the videos using the Dyadic Mini Code, which includes six categories: mutual attention, positive affect, turn-taking, parental pauses, infant cues, and parental sensitive responsiveness. Scores range from 6 to 12, with ≥10 indicating synchronous interaction.
Parent-infant interaction | GW 32 +/- 2 weeks
  All three diaper changes will be video recorded with both parents present and instructed to act as they normally would. Parent sensitivity towards the infant will be assessed from the videos using Ainsworth's Sensitivity Scales. This instrument constitutes of four sub-scales measuring sensitivity, cooperation, availability and acceptance. Each scale range 1-9, where higher scores indicate better interactive behaviour.

SECONDARY OUTCOMES:
Skin temperature in mother, father and infant | GW 32 +/- 2 weeks
  Correlation of skin temperature in the triad will be measured at the forehead on infants and both parents before and after each diaper change with an infrared thermometer. This method is painless as the temperature can be assessed without touching the infant.
Infant development | 6 and 12 months corrected age, +/-2 months
  The Swedish Ages and Stages Questionnaire: Social Emotional (ASQSE2) is a 25-item tool assessing children's social-emotional development.
Infant temperament | 6 and 12 months corrected age, +/-2 months
  Infant Behaviour Questionnaire-Revised short form, which assesses infants' temperament across three main components (negative emotionality, positive affectivity/surgency, and orienting/regulatory capacity), will be administered when infants are 6 and 12 months corrected age. This questionnaire includes 14 scales measured on 7-point-scales. A min-max score for each scale is 1-7 where 7 indicates a higher frequency of the specific behaviours being measured.
Communicative Skills and Language Abilities | 12 months corrected age, +/-2 months
  The Early Communicative Development Inventories (words & gestures), assess communicative skills and language abilities of infants aged 8-16 months. The Swedish version will be used to evaluate the child's understanding of words, vocabulary, and communicative gestures. Confirmative answers are given in a form of examples.

OTHER OUTCOMES:
Parental-to-infant emotional bonding | GW 32 +/- 2 weeks
  The Swedish version of the Mother-to-Infant-Bonding-Scale (MIBS), which assesses parental emotions toward their infants over the past ten days using a 4-point Likert scale ranging 0-3. Higher scores indicate more bonding challenges.
Parental postpartum depression | GW 32 +/- 2 weeks
  The well-established Edinburgh Postnatal Depression Scale (EPDS, a ten-item questionnaire scoring symptoms of depression in new parents over the past week on a scale ranging from 0 to 3, higher scores indicating more symptoms of depression.
Parental well-being | GW 32 +/- 2 weeks
  World Health Organization-5 (WHO-5), comprising six questions measuring well-being on a scale of 0-5 points scale, with scores translated to a percentage where 100% indicates maximum well-being.
Parental anxiety | GW 32 +/- 2 weeks
  Spielberger's Anxiety Inventory-State short version has six questions measuring anxiety (right now) on a 4-point likert scale. Total scores range from 6-24, higher scores indicate more anxiety.
Experinces of connection with baby | GW 32 +/- 2 weeks
  Each parent will be asked to write a narrative about their own feelings of connection to the baby in relation to the diaper change and in general.
Parental distress | When the infant is 6 and 12 months +/-2 months
  The Distress Thermometer-Parent (DT-P), designed to identify parent distress over the past week using a visual Likert-scale thermometer ranging from 0 to 10 points where higher scores indicate more distress. Additionally, parents indicate 'yes' or 'no' to a problem list encompassing practical, social, emotional, physical, cognitive, and parenting issues, elucidating the source of distress.

CONTACTS AND LOCATIONS:
Locations (1):
- H.R.H Crown Princess Victoria's Children's and Youth Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided